CLINICAL TRIAL: NCT06703853
Title: Identifying Tissue-of-origin and Gene Expression Program by Immunoprecipitation of Cell-free Nucleosomes in Transplant Patients and Patients with Malignancies.
Brief Title: Identifying Tissue-of-origin in Transplant Patients and Patients with Malignancies.
Acronym: cfDNA
Status: Active, not recruiting | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, Eithan Galun, Principal Investigator, Hadassah Medical Organization
Other Study IDs: 0030-19-HMO; Israel ministry of health (Other: Israel ministry of health)
Record Dates: First submitted 2024-11-12; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-07

CONDITIONS: Malignancies
Keywords: gene expression; DNA; Liver cancer
MeSH Terms: conditions — Neoplasms; Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and urine samples for cfDNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
the investigators are developing a method for diagnosing cell death in the body using blood and urine tests. The test is based on two well-known phenomena in biology. First, when cells in the body die, short fragments of their DNA, about 150 bases long, find their way into the bloodstream for a short period of time of about fifteen minutes to an hour, before being eliminated in the liver and kidney. The details of this process are not fully known, but it is clear that the phenomenon exists. Already today, this phenomenon is widely used clinically for prenatal diagnosis of chromosomal aberrations in the DNA of the fetus that is found in large quantities in the mother's blood. Liquid biopsies from cancer have already been developed, based on the identification of somatic mutations originating from a cancerous tumor in the free DNA found in the serum or plasma. In the case of cancer, liquid biopsies may be a convenient way to monitor the genetic evolution of the tumor, response to treatments, and more. This approach of detecting cell death using free DNA in the bloodstream has a severe limitation when it comes to the death of cells whose genome is not different from the genome of the other tissues in the body, and therefore the DNA cannot be associated with the tissue of origin based on sequence analysis.

DETAILED DESCRIPTION:
The duration of the sample collection period is estimated to be five years. Work in the laboratory will continue for another 3 years. The laboratory work will be carried out in the laboratories of Prof. Eithan Galun at Hadassah Ein Kerem and Prof. Nir Friedman at the Hebrew University of Givat Ram. Access will be given to Prof. Galun and his team. Since genetic variation is not tested in this study, there is no fear of revealing the subject's personal genetic information. In this study we use an identified sample, on which identifying details for the participant are indicated, for example: name, social security number or code number that can be given to the sample. The identified information and the information that will be extracted from the sample will be saved in coded excel sheets. In this way, only authorized researchers and research staff will be allowed access. The samples will be preserved as coded identified samples in the laboratory of Prof. Eithan Galun, Hadassah Ein Kerem, Jerusalem in a freezer in a locked room with limited access to researchers and the authorized research team only, and also, in the laboratory of Prof. Nir Friedman, the Hebrew University of Givat Ram, Jerusalem under similar conditions with access to the research team only. the investigators also ask the liver and kidney transplant recipients to collect a urine sample, with the thought that it might be possible to save a blood test and be satisfied with a urine sample.

ELIGIBILITY:
Inclusion Criteria:

Kidney and liver transplant recipients Patients with malignant tumors

Exclusion Criteria:

Pregnant women Minors Incompetent Chronic background disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney and liver transplant recipients
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-12 (Estimated)

PRIMARY OUTCOMES:
Improvement of liver function tests including ALT and AST levels after immunosuppression | Measurements of liver enzymes after diagnosis of acute rejection
  Reduction of liver enzymes following immunosuppression treatment

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Hamburger, MRS, Study Chair — Gene Therapy Institute
Locations (1):
- Hdassah Hospital, Jerusalem, Israel

IPD SHARING:
Plan to Share IPD: Yes
Publication
Supporting Information: Study Protocol
Time Frame: January 2028 for 7 years.
Access Criteria: After publication any one.
URL: https://www.eithangalun.com/